CLINICAL TRIAL: NCT04373577
Title: Comparison of Ultrasound Guided Erector Spinae Plane Block and Ultrasound Guided Pericapsular Nerve Group Block for Pediatric Hip Surgery
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Tanta University (Other)
Responsible Party: Principal Investigator, tarek abdel hay mostafa, principle investigator, Tanta University
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Supportive Care
Other Study IDs: ESP block and PENG block
Record Dates: First submitted 2020-04-28; First posted 2020-05-04 (Actual); Last update posted 2022-11-25 (Actual); Status verified 2022-11

CONDITIONS: Postoperative Pain
MeSH Terms: conditions — Pain, Postoperative

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- ESP group (Experimental): Under ultrasound guidance, patients of this group will receive (0.5ml/kg) plain bupivacaine 0.25%with adrenaline 2.5 µg/ml injected beneath the erector spinae muscle sheath at the level of the transverse process of the second lumbar vertebrae
  Interventions: Procedure: erector spinae plane block
- PENG group (Experimental): Under ultrasound guidance, patients of this group will receive (0.5ml/kg) plain bupivacaine 0.25%with adrenaline 2.5 µg/ml injected as the tip of the needle in the musculofascial plane between the psoas tendon anteriorly and the pubic ramus posteriorly
  Interventions: Procedure: pericapsular nerve group block

INTERVENTIONS:
Procedure: erector spinae plane block — the patient will be placed in the lateral position with the surgical side up for performing erector spinae plane block. After skin preparation, superficial (5-12 MHz) ultrasound transducer will be placed in a longitudinal orientation 1-2cm lateral to the midline at the sacral level. The L2 level will be identiﬁed by counting upward from the sacrum. Following identiﬁcation of the erector spinae muscle (ESM) and transverse process, a 21 G needle will be inserted deep to the erector spinae muscle (ESM) in a cranio-caudal direction. After negative aspiration, the correct needle position will be conﬁrmed with the administration of 0.5-1ml LA. A total volume of 0.5 mL/kg local anesthetic solution will be injected interfascial plane between erector spinae muscle and transverse process for block performance.
  Arms: ESP group
Procedure: pericapsular nerve group block — the patient will be in supine position. The ilio-pubic eminence (IPE), the iliopsoas muscle and tendon, the femoral artery, and pectineus muscle will be visualized using a linear ultrasound probe. A 22-gauge, 50-mm needle will be introduced in a lateral to medial fashion in an in-plane approach to place the tip of the needle in the musculofascial plane between the psoas tendon anteriorly and the pubic ramus posteriorly. Following negative aspiration, a total volume of 0.5 mL/kg local anesthetic solution will be injected.
  Arms: PENG group

SUMMARY:
Surgical repair of the hip can be extremely painful and is associated with considerable postoperative pain in children despite the use of systemic opioids. These patients may benefit from neuraxial analgesia in adjunction with general anesthesia. The reported advantages of this technique include decreased opiate exposure, decreased time in the post-anesthesia recovery room, decreased hospital stay, reduce the post-operative morbidity, provide early mobilization. Regional anesthetic techniques seem to be a better choice for improving acute pain management in these patients, with fewer adverse effects.

DETAILED DESCRIPTION:
Surgical repair of the hip can be extremely painful and is associated with considerable postoperative pain in children despite the use of systemic opioids. These patients may benefit from neuraxial analgesia in adjunction with general anesthesia. The reported advantages of this technique include decreased opiate exposure, decreased time in the post-anesthesia recovery room, decreased hospital stay, reduce the post-operative morbidity, provide early mobilization.

Regional anesthetic techniques seem to be a better choice for improving acute pain management in these patients, with fewer adverse effects. The erector spinae block is a recently described ultrasound-guided technique in which local anesthetics is injected into a fascial plane between the tips of the thoracic transverse processes and the overlying erector spinae muscle (longissimus thoracis).

Pericapsular nerve group (PENG) block has been recently recommended by Girón-Arango et al. for use as postoperative analgesia in hip surgeries. It is a new regional anesthesia technique in the region between the anterior inferior iliac spine (AIIS) and ilio-pubic eminence (IPE).

The anterior capsule is the most richly innervated section of the joint suggesting these nerves should be the main targets for hip analgesia.

ELIGIBILITY:
Inclusion Criteria:

* Children of both genders
* American Society of Anaestheologists (ASA) physical activity I, II
* aged more than one year
* admitted for elective pediatric hip surgery

Exclusion Criteria:

* Children with severe systemic disease with American Society of Anaestheologists (ASA) III or IV,
* children with previous neurological or spinal disorders,
* coagulation disorder,
* infection at the block injection site,
* history of allergy to local anesthetics
* bilateral hip surgery.

Ages: 1 Year to 6 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 56 (Actual)
Dates: Start 2020-05-01 (Actual); Primary Completion 2022-09-01 (Actual); Study Completion 2022-10-01 (Actual)

PRIMARY OUTCOMES:
Time to first rescue analgesic demand | postoperative first day
  Time to first rescue analgesic requirement: measured from the end of surgery till patient require analgesia.

SECONDARY OUTCOMES:
Total doses of intraoperative fentanyl consumption | intraoperative
  Total doses of intraoperative fentanyl consumption
Total analgesic consumption | postoperative first day
  Total analgesic consumption If pain score more than 3, the child will be given intravenous morphine as rescue analgesia will be given in a dose 0.1mg/kg.

CONTACTS AND LOCATIONS:
Locations (1):
- Tarek Abdel Hay, Tanta, El Gharbyia, Egypt